CLINICAL TRIAL: NCT05460546
Title: A Multicenter, Randomized, Double-blind, Dose-parallel, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of Jincaopian Tablets in Subjects With Chronic Pelvic Pain After Pelvic Inflammatory Disease
Brief Title: The Effect of Jincaopian Tablets on Chronic Pelvic Pain After Pelvic Inflammatory Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z-JCP-T-II-2020-HMZC-01
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jincaopian Tablets high-dose group (Experimental): Patients receive high dose Jincaopian Tablets 0.6g/day for 12 weeks.
  Interventions: Drug: Jincaopian Tablets high dose
- Jincaopian Tablets low-dose group (Experimental): Patients receive low dose Jincaopian Tablets 0.3g/day for 12 weeks.
  Interventions: Drug: Jincaopian Tablets low dose
- Placebo group (Placebo Comparator): Patients receive a matching placebo for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Jincaopian Tablets high dose — Jincaopian Tablets 0.2g tid p.o.
  Other Names: ZY5301
  Arms: Jincaopian Tablets high-dose group
Drug: Jincaopian Tablets low dose — Jincaopian Tablets 0.1g tid p.o.
  Other Names: ZY5301
  Arms: Jincaopian Tablets low-dose group
Other: Placebo — Placebo tid p.o.
  Arms: Placebo group

SUMMARY:
This phase II trial attempts to evaluate the efficacy and safety of Jincaopian Tablets in the treatment of subjects with chronic pelvic pain after pelvic inflammatory disease.

DETAILED DESCRIPTION:
Chronic pelvic pain is the major sequela of pelvic inflammatory disease and it's a common, burdensome, and costly condition that disproportionately affects women. This multicenter, randomized, double-blind, dose-parallel, placebo-controlled phase II clinical trial is designed to evaluate the efficacy and safety of Jincaopian Tablets in the treatment of subjects with chronic pelvic pain after pelvic inflammatory disease. In this trial, 180 subjects were enrolled and randomized to either "high-dose Jincaopian Tablets" group, "low-dose Jincaopian Tablets " group, or the "placebo" group in a 1:1:1 ratio. The treatment period is 12 weeks and the follow-up period is 4 weeks. The outcome measures of chronic pelvic pain relief in this trial are pain visual analog scale (VAS), modified McCormick scale and SF-12 Score.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for chronic pelvic pain sequelae of pelvic inflammatory disease;
* The average VAS score of pain in the week before enrollment is ≥4;
* The McCormack scale of physical signs at the time of enrollment is 4 to 12 points (including 4 points and 12 points);
* Women aged 18 to 55 (including 18 and 55) with a history of sexual life;
* Voluntarily participate in this clinical trial, give informed consent and sign the informed consent form.

Exclusion Criteria:

* Pelvic inflammatory disease (acute attack);
* Pregnant or lactating women, women of childbearing age who are unwilling to take effective measures to prevent pregnancy during the trial and within 3 months after the trial;
* Critically ill or with surgical indications;
* Previously diagnosed with cervical intraepithelial neoplasia, primary/secondary dysmenorrhea, pelvic stasis syndrome and chronic pelvic pain caused by other non-pelvic inflammatory diseases;
* Complicated with specific vaginitis such as vulvovaginal candidiasis, trichomonas vaginitis, bacterial vaginosis, etc.;
* Gynecological tumors (maximum diameter of uterine fibroids greater than 3cm and submucosal fibroids), endometriosis, adenomyosis, acute cervicitis, tuberculous pelvic inflammatory disease, interstitial cystitis and other diseases related symptoms;
* Placement of intrauterine device in the past 3 months; absence of uterus and bilateral appendages;
* Received related treatment or took drugs with similar functions and indications within 14 days before the introduction;
* Have a history of allergy to the components of the test drug;
* Participated in other clinical trials within the past 3 months;
* The investigator believes that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale (VAS) | Baseline to 16 weeks
  To measure patient's pain intensity (most commonly) along a 100 mm horizontal line daily.
Modified McCormick Scale | Baseline and at Weeks 4, 8, 12, 16
  To evaluate the total score of the physical sign scale and the scores of each part including abdominal tenderness, rebound tenderness, and gynecological examination compared with the baseline in each group at weeks 4, 8, 12, 16.
SF-12 Score | Baseline and at Weeks 12
  To evaluate the health status of the patients compared with the baseline in each group at weeks 12.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuxiang Teng, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Teng X, Li H, Yang D, Gao Z, Cui L, Chen H, Song Q, Xu L, Li H, Zhang Q, Wu J, Leng J. ZY5301 Tablet vs Placebo for Treatment of Chronic Pelvic Pain After Pelvic Inflammatory Disease: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2423229. doi: 10.1001/jamanetworkopen.2024.23229. PMID 39042407